CLINICAL TRIAL: NCT00490126
Title: Data Collection of Demographics and Perioperative Care of Patients Undergoing Laparoscopic Surgery in the Department of Gynecologic Oncology
Brief Title: Data Collection of Demographics and Perioperative Care of Patients Undergoing Laparoscopic Surgery
Status: Terminated | Type: Observational
Why Stopped: Not enough staff
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2006-0170
Record Dates: First submitted 2007-06-20; First posted 2007-06-22 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Laparoscopy
Keywords: Laparoscopic Surgery; Laparoscopy; Gynecology; Demographics; Perioperative Care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Laparoscopic Surgery Database
  Interventions: Other: Laparoscopic Surgery Data Collection

INTERVENTIONS:
Other: Laparoscopic Surgery Data Collection — Prospectively and retrospectively collect data on patients who had laparoscopic surgery since January 1, 1990 forward. Data from the initial patient visit note, consultation notes, operative report, discharge summary, and follow-up progress notes will be entered into the database.

SUMMARY:
The goal of this clinical research study is to collect information on patients who had or are going to have laparoscopy performed at M. D. Anderson. Researchers want to use this information to learn the effects of laparoscopic surgery on patients over time.

DETAILED DESCRIPTION:
If you agree to take part in this study, your demographic information (such as your age, race, medical and surgical history, and type of cancer) will be collected. Information about the type of surgical procedure performed on you, your care during and after your surgery, any problems related to your surgery, and details about your follow-up care will be entered into a research database. This information will be collected from patients seen at M. D. Anderson since January 1, 1990. It will be used for future research studies.

The research database will be updated, after about 1 year, to include information on your disease outcome, treatment, and/or follow-up care. This information will be collected from your medical record, if possible. If it is not in your medical record, you may again be contacted so that researchers can learn this information.

Your participation in this study will continue up to 5 years after your laparoscopic procedure.

This is an investigational study. Up to 1,000 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. All patients who had or will have laparoscopic surgery in the Department of Gynecologic Oncology (Gynecologic Oncology and General Gynecology) since January 1, 1990 forward.

Exclusion Criteria: None

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who had or will have laparoscopic surgery in the Department of Gynecologic Oncology (Gynecologic Oncology and General Gynecology) since January 1, 1990 forward.
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2006-06-15 (Actual); Primary Completion 2018-09-18 (Actual); Study Completion 2018-09-18 (Actual)

PRIMARY OUTCOMES:
Collect, both prospectively and retrospectively, data on demographics, perioperative care, and patient outcomes in patients undergoing laparoscopic surgery. | 21 Years

SECONDARY OUTCOMES:
Organize clinical information, patient characteristics, treatment, and laparoscopic outcome data into a single data repository, maintained in a secure platform that will provide an archive for future research. | 21 Years

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Ramirez, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org